CLINICAL TRIAL: NCT04658446
Title: Comparison Between Augmented Reality-Assisted Bonding Versus Digitally-Assisted Indirect Bonding in Orthodontic Patients (Randomized Clinical Trial)
Brief Title: Augmented Reality-Assisted Bonding Versus Digitally-Assisted Indirect Bonding in Orthodontic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seif El-Din Amr Hussein Hegab (Other)
Responsible Party: Sponsor-Investigator, Seif El-Din Amr Hussein Hegab, PhD Candidate/ Researcher, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: ORTH 3-3-2
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Augmented Reality
Keywords: Augmented Reality; Indirect Bonding; Digital Orthodontics; Orthodontic bracket

STUDY DESIGN:
Intervention Model Description: 8 Patients with Split-mouth trial design. Full permanent dentition. In need of Orthodontic treatment with fixed appliance therapy.
Who Masked: Outcomes Assessor
Masking Description: The assessor shall not know which group is which in the accuracy outcome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Reality-Assisted Bonding (Experimental): The quadrant of the upper arch that shall use the AR-assisted bonding method. From the maxillary central incisor to the maxillary first permanent molar of the same quadrant.
  Interventions: Device: Augmented Reality-Assisted Indirect Bonding
- Digitally-Asssited Indirect Bonding (Active Comparator): The quadrant of the upper arch that shall use the digitally-assisted bonding method utilizing a 3D printed tray. From the maxillary central incisor to the maxillary first permanent molar of the same quadrant.
  Interventions: Device: Digitally-Asssited Indirect Bonding

INTERVENTIONS:
Device: Augmented Reality-Assisted Indirect Bonding — Virtual Orthodontic attachments are overlaid on top of the patient's teeth using an augmented-reality headset to guide the bracket positioning procedure.
  Arms: Augmented Reality-Assisted Bonding
Device: Digitally-Asssited Indirect Bonding — 3D printed models with precise brackets positioned as virtually pre-planned. To aid in the transfer of the planned bracket positions to the patient's physical teeth.
  Other Names: 3D Printed Indirect Bonding Guides
  Arms: Digitally-Asssited Indirect Bonding

SUMMARY:
Comparing two indirect bonding techniques. Augmented Reality-assisted bonding and Digital 3D printed indirect bonding trays in regards to patient convenience, accuracy of bracket placement and time consumption of each technique used.

DETAILED DESCRIPTION:
Augmented reality is a relatively new addition to the digital armamentarium. It is becoming increasingly popular especially among surgeons, whether general or dental. In light of the clinicians whom have relied on augmented reality in their fields of work, it was suggested that an augmented reality-assisted orthodontic bonding guide be of use. Such an application would theoretically solve many issues of the indirect bonding techniques at hand.

In this study, we shall investigate whether the theory behind such an augmented reality-assisted bonding guide is on par with the digitally-assisted indirect bonding in terms of patient convenience, accuracy of bracket placement and time consumption of the bonding process, to see whether it qualifies to be a method among all the other methods stated in the literature for indirect bonding.

Digital indirect bonding has many advantages, one of which is achieving greater accuracy in bracket positioning, however it has some down sides such as excess composite flashes around brackets after curing and the cost of 3D printing.

Aim of the Study Is to evaluate the patients' convenience upon using the newly introduced augmented reality-assisted bonding guide in comparison to the digitally-assisted indirect bonding tray. Secondary objectives such as accuracy and procedure time consumption between the two methods are also of importance.

Null Hypothesis There will be no difference in the patients' convenience, accuracy and procedure time consumption between the two methods proposed.

Trial Design Split-mouth, randomized, clinical superiority trial with 1:1 allocation ratio.

Sample Size 96 Teeth with different attachments (Brackets and Tubes)

ELIGIBILITY:
Inclusion Criteria:

* Arch length deficiency ≤ 5 mm.
* Good oral hygiene.
* Fully erupted permanent dentition, not necessarily including third molars.

Exclusion Criteria:

* Patient with active periodontal diseases.
* Anterior cross-bite.
* Enamel hypoplasia.
* Previous orthodontic treatment.
* Teeth with caries or restorations on labial surfaces.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-02-25 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-25 (Estimated)

PRIMARY OUTCOMES:
Patient Convenience | Immediately after the bonding procedure.
  Whether the patient was at ease during the bonding procedure or not and the overall convenience of the procedure from the patient's point of view.

SECONDARY OUTCOMES:
Accuracy of the Method | After one week of the Bonding Procedure.
  Whether the bracket positions were identical to the virtually-planned positions or not. Measured using specialized software for superimposing two 3D virtual models and measuring the differences.
Time | At the time of the Bonding Procedure.
  The actual time consumed to bond all attachments using both techniques. This shall include Lab-time and Chair-side time.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Castilla AE, Crowe JJ, Moses JR, Wang M, Ferracane JL, Covell DA Jr. Measurement and comparison of bracket transfer accuracy of five indirect bonding techniques. Angle Orthod. 2014 Jul;84(4):607-14. doi: 10.2319/070113-484.1. Epub 2014 Feb 20. PMID 24555689
- [Result] El-Timamy AM, El-Sharaby FA, Eid FH, Mostafa YA. Three-dimensional imaging for indirect-direct bonding. Am J Orthod Dentofacial Orthop. 2016 Jun;149(6):928-31. doi: 10.1016/j.ajodo.2015.12.009. PMID 27242004
- [Result] Kwon HB, Park YS, Han JS. Augmented reality in dentistry: a current perspective. Acta Odontol Scand. 2018 Oct;76(7):497-503. doi: 10.1080/00016357.2018.1441437. Epub 2018 Feb 21. PMID 29465283